CLINICAL TRIAL: NCT03582618
Title: A Phase 2, Open-Label Study With Orally Administered CVM-1118 and Sorafenib in Subjects With Advanced Hepatocellular Carcinoma
Brief Title: CVM-1118 and Sorafenib Combination in Subjects With Advanced Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study has been terminated due to slow enrollment
Sponsor: TaiRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVM-004
Record Dates: First submitted 2018-05-21; First posted 2018-07-11 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma; Advanced Cancer
Keywords: Oncology; Hepatocellular Carcinoma (HCC); Sorafenib; Hepatoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sorafenib + CVM-1118 (Experimental): Cycle 0 (at least 3 weeks): sorafenib tolerability assessment period (sorafenib alone)
  400mg BID daily (starting dose); The subject will be assessed for the need for a dose reduction in sorafenib during this period.
  Cycle 1+ (28-day cycles): combination period (sorafenib+CVM-1118)
  Tolerable dose of sorafenib and CVM-1118 150 (starting dose) or 200 mg BID will be administered continuously for a 28-day cycle until progressive disease, unacceptable toxicity, or consent withdrawal.
  Interventions: Drug: Sorafenib; Drug: CVM-1118

INTERVENTIONS:
Drug: Sorafenib — Sorafenib will be administered orally at a starting dose of 400mg BID daily and the necessity of dose reduction will be assessed during sorafenib tolerability assessment period
  Other Names: Nexavar
Drug: CVM-1118 — CVM-1118 will be administered orally at 150 mg BID or 200 mg BID daily and combined with the tolerable dose of sorafenib for a 28-day cycle
  Other Names: TRX-818

SUMMARY:
CVM-1118 is a new small molecule chemical entity being developed as a potential anti-cancer therapeutic by TaiRx, Inc. CVM-1118 is a potent anti-cancer agent in numerous human cancer cell lines. The safety of administrating CVM-1118 on human is evaluated from the phase 1 study. The objectives of the phase 2 study is to further investigate the efficacy of CVM-1118 with sorafenib for subjects with advanced hepatoma.

DETAILED DESCRIPTION:
Sorafenib is a multi-kinase inhibitor that inhibits tumor growth and angiogenesis. Although sorafenib is the first-line treatment of advanced hepatocellular cancer (HCC), patients developing resistance to sorafenib have been reported.

To meet the medical need, TaiRx, Inc. develops a new small molecule drug, CVM-1118 targeting the formation of vasculogenic mimicry (VM). VM has been associated with tumor metastasis and poor clinical outcomes. VM is reported to be particularly active in tumor under hypoxia state when patients are treated with the potent vascular endothelial growth factor (VEGF) inhibitor like sorafenib. Hence, the ability of inhibiting the VM network make CVM-1118 a potential good combination drug with sorafenib for advanced diseases.

The safety profile of CVM-1118 dosing has been established in the phase 1 study. The analysis of metabolism pathways further showed that the potential of CVM-1118 and sorafenib drug-drug interactions are very low.

Based on the mechanism of actions and the safety analysis of sorafenib and CVM-1118, the design of phase 2 trial with the combination therapy might have great potential for the patients with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, informed consent
2. Age 18 or older (for all treatment locations with exception of Taiwan), or age 20 or older (Taiwan only)
3. Pathologically or cytologically-confirmed, advanced-stage hepatocellular carcinoma without prior systemic treatment except for prior immunotherapy and Child-Pugh liver function class A appropriate for treatment with sorafenib
4. Measurable disease according to modified Response Evaluation Criteria in Solid Tumors criteria (mRECIST)
5. Eastern Cooperative Oncology Group (ECOG) performance status: 0 to 1
6. Adequate laboratory parameters including:

   1. Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 3.0 x upper limit of normal (ULN), or AST and ALT ≤ 5.0 x ULN if liver function abnormalities are due to underlying malignancy
   2. Total serum bilirubin ≤ 2.0 x ULN (except for subjects with documented Gilbert's syndrome who have a limit of ≤ 3.0 x ULN)
   3. Absolute neutrophil count (ANC):1500/µL
   4. Platelets: 90,000/µL
   5. Hemoglobin: 9.0 g/dL
   6. Serum creatinine ≤ 2.0 x ULN or creatinine clearance of ≥ 50 mL/min
   7. Serum albumin ≥ 3.0 g/dL
   8. International normalized ratio (INR) ≤ 1.4
   9. Prothrombin Time (PT)/ Activated Partial Thromboplastin Time (aPTT) ≤ 1.2 x ULN
7. QTc interval (using Fridericia correction) of ≤ 470 msec (QTc interval may be derived from up to 3 separate EKGs performed at least 5 minutes apart)
8. Willingness to participate in collection of pharmacokinetic and other exploratory blood collection as defined in the protocol
9. Willingness to use adequate contraception throughout study and for a period of 3 months after last dose of CVM-1118

Exclusion Criteria:

1. Major surgery (other than diagnostic surgery) or radiation therapy within 28 days of starting study treatment
2. Prior systemic immunotherapy for hepatoma within 28 days of starting study treatment
3. Systemic anticancer therapy (e.g., chemotherapy, hormonal, investigational, biological therapies) within 28 days (or fewer than 5 half-lives, whichever is shorter) of starting study treatment except for ongoing hormonal therapy administered for control of a second cancer (e.g., breast or prostate cancer)
4. Receipt of a CYP3A4 inducer less than 28 days or 5 half-lives of the CYP3A4 inducer prior to the first day of sorafenib administration
5. Other known active cancer(s) likely to require treatment in the next two (2) years or likely to impact the assessment of any study endpoints
6. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy (e.g., subjects with known HBV or HCV infections controlled on antivirals are allowed)
7. Known Central Nervous system (CNS) metastases unless appropriately treated and neurologically stable for ≥ 4 weeks off steroids
8. Pregnant or currently breast-feeding
9. Known HIV-positive
10. Patients with impaired gastrointestinal (GI) diseases that may significantly alter the absorption of oral medications
11. Psychiatric illness/social situations that would interfere with compliance with study requirements
12. History of clinically significant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure (New York Heart Association classification ≥ 2), unstable angina, poorly controlled arrhythmias, myocardial infarction within 6 months of study entry
13. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that would impart, in the judgement of the PI and/or Sponsor, excess risk associated with study participation or study drug administration, which would make the subject inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24 weeks after the last subject starts CVM-1118
  Assessment by modified RECIST criteria

SECONDARY OUTCOMES:
Overall survival (OS) | 24 weeks after the last subject starts CVM-1118 and up to 1 year after the last-dose
  Overall survival (OS) is defined as time from first dose of study drug to death
Progression-free survival (PFS) | 24 weeks after the last subject starts CVM-1118 and up to 1 year after the last-dose
  Progression-free survival (PFS) is defined as time from the first dose of study drug to the time of progression or death
Time to progression (TTP) | 24 weeks after the last subject starts CVM-1118 and up to 1 year after the last-dose
  Time to progression (TTP) is defined as the time from the first dose of study drug to the time of progression
Duration of response (DoR) | 24 weeks after the last subject starts CVM-1118 and up to 1 year after the last-dose
  Duration of response (DoR) is defined as time from the first documentation of response to the time of progression
Disease control rate (DCR) | 24 weeks after the last subject starts CVM-1118 and up to 1 year after the last-dose
  Disease control rate (DCR) is defined as the sum of complete response (CR), partial response (PR), and stable disease rate (SD) as assessed by modified RECIST criteria
Rate of Adverse event (AE) and Serious Adverse Event (SAE) | During the course of trial and within 28 days following the last dose of CVM-1118 or prior to the start of new treatment, whichever comes first
  Rate of Adverse event (AE) and Serious Adverse Event (SAE) are assessed using Common Terminology Criteria for Adverse Events v5 (CTCAE) criteria
Assessed the baseline and out-of-range vital signs_ body temperature, blood pressure, heart rate, and respiratory rate by CTCAE v4.03 | During the course of trial and within 28 days following the last dose of CVM-1118 or prior to the start of new treatment, whichever comes first
  A list of all laboratory normal ranges will also be provided. Values with CTCAE v4.03 Grade ≧ 3 will be identified with flags.
Assessed the baseline and out-of range laboratory parameters_hematology, chemistry, coagulation, and urinalysis by CTCAE v4.03 | During the course of trial and within 28 days following the last dose of CVM-1118 or prior to the start of new treatment, whichever comes first
  A list of all laboratory normal ranges will also be provided. Values with CTCAE v4.03 Grade ≧ 3 will be identified with flags.
Abnormalities in electrocardiography (ECG) | During the course of trial and within 28 days following the last dose of CVM-1118 or prior to the start of new treatment, whichever comes first
  a 12-lead (with a 10-second rhythm strip) tracing, with a capacity to calculate the standard intervals automatically, will be used.
Maximum Plasma Concentration [Cmax] of sorafenib, CVM-1118, and its metabolite CVM-1125 after CVM-1118 dosing | During Cycle 1 and Cycle 2 (each cycle is 28 days)
  Maximum Plasma Concentration [Cmax] of sorafenib, CVM-1118, and its metabolite CVM-1125 will be measured to see maximum exposure after CVM-1118 dosing
Area Under the Curve [AUC] of sorafenib, CVM-1118, and its metabolite CVM-1125 after CVM-1118 dosing | During Cycle 1 and Cycle 2 (each cycle is 28 days)
  Area Under the Curve [AUC] of sorafenib, CVM-1118, and its metabolite CVM-1125 will be measured to see drug exposure after CVM-1118 dosing
Pharmacodynamics analysis for the relationship of Cmax and ORR | During Cycle 1 and Cycle 2 (each cycle is 28 days)
  Relationship between Cmax and ORR will be evaluated
Pharmacodynamics analysis for the relationship of AUC and ORR | During Cycle 1 and Cycle 2 (each cycle is 28 days)
  Relationship between AUC and ORR will be evaluated
Pharmacodynamics analysis for the relationship of Cmax and Adverse Event (AE) | During Cycle 1 and Cycle 2 (each cycle is 28 days)
  Relationship between Cmax and AE will be evaluated
Pharmacodynamics analysis for the relationship of AUC and Adverse Event (AE) | During Cycle 1 and Cycle 2 (each cycle is 28 days)
  Relationship between AUC and AE will be evaluated

CONTACTS AND LOCATIONS:
Locations (3):
- Charleston Hematology Oncology Associates, Charleston, South Carolina, United States
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei